CLINICAL TRIAL: NCT00620607
Title: A Phase II, Open Label, Multiple Center Study of huC242-DM4 Given as an Intravenous Infusion Once Every Three Weeks to Patients With Metastatic Gastric or Gastroesophageal Junction Carcinomas
Brief Title: huC242-DM4 Treating Patients With Metastatic Gastric or Gastroesophageal Junction Carcinomas
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of accrual
Sponsor: ImmunoGen, Inc. (Industry)
Responsible Party: Clinical Operations, ImmunoGen, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMGN 102
Record Dates: First submitted 2008-02-07; First posted 2008-02-21 (Estimated); Last update posted 2015-08-26 (Estimated); Status verified 2009-04

CONDITIONS: Stomach Neoplasms; Metastatic or Locally Advanced Gastric Cancer; Metastatic or Local Advanced GE Junction Cancer
Keywords: gastric
MeSH Terms: conditions — Stomach Neoplasms; Neoplasm Metastasis

INTERVENTIONS:
Drug: huC242-DM4 — dose of 126 mg/m2 or 168 mg/m2 given as IV once every 3 weeks

SUMMARY:
To assess the response rate of huC242-DM4 given as an intravenous infusion to patients with metastatic or locally advanced gastric or gastroesophageal junction cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients must understand and voluntarily sign an informed consent.
* Patients must have histological documentation of metastatic or locally advanced (American Joint Committee on Cancer Staging System: Stages IIIA, IIIB, and IV) gastric or gastroesophageal junction adenocarcinoma.
* Patients must have ECOG performance status < 1.
* Patients must be at least 18 years of age.
* Patients who have been treated with only one prior chemotherapy regimen and who have documented disease progression.
* Patients must have confirmation of CanAg expression performed prior to enrollment by immunohistochemical assessment for CanAg on archived biopsy samples.
* Patients must have measurable disease with at least one lesion that can be accurately measured by Response Evaluation Criteria in Solid Tumors (RECIST). The lesion size must be at least 20 mm by conventional radiological techniques or at least 10 mm by spiral CT scan. Disease in an irradiated field as the only site of measurable disease is acceptable if there has been a clear progression of the lesion.
* Patients with reproductive potential must agree to use an effective contraceptive method during the study and for 30 days after receiving the last dose of study drug.
* Women of childbearing potential (WCBP) must have a negative urine or serum pregnancy test within one week prior to enrollment in the study.
* Patients must have any chemotherapy, immunotherapy, hormonal therapy, radiotherapy for cancer or surgery (except for minor surgical procedures) completed at least 3 weeks before starting study medication.
* Patients must have resolution of all clinically significant toxic effects (excluding alopecia) of any prior treatments including surgery, radiotherapy, hormone therapy, immunotherapy, targeted non-cytotoxic therapy, or chemotherapy to grade ≤ 1 by NCI CTCAE v. 3.0 unless otherwise specified in the inclusion laboratory values.
* Patients must have adequate organ function including:

  1. Hematopoietic:

     i. Absolute neutrophil count > 1,500/mm3. ii. Platelet count > 100,000/mm3. iii. Hemoglobin > 9 g/dL (transfusion allowed).
  2. Renal:

     i. Serum creatinine ≤ 1.5 x the upper limit of normal (ULN) ii. Calculated creatinine clearance > 60 mL/min/1.73m2.
  3. Hepatic:

     i. Alanine aminotransferase (ALT), or aspartate aminotransferase (AST) ≤ 2.5 x ULN ii. Total bilirubin ≤ 1.5 x ULN

     Exclusion Criteria:
* Pregnant or lactating women. Women of childbearing potential (WCBP) must have a negative urine or blood test for pregnancy before first treatment.
* Known hypersensitivity to previous monoclonal antibody therapy or maytansinoids.
* Active and uncontrolled infection.
* Known history hepatitis B or C, HIV, or history of alcoholic liver disease.
* Patients with any serious medical or psychiatric disorder that would interfere with patient safety or informed consent.
* Patients with peripheral neuropathy grade 2 or greater.
* Patients with known leptomeningeal disease or progressive brain metastasis. Routine screening with CNS imaging studies (CT or MRI) is required only if clinically indicated.
* Patients with concomitant malignancies or previous malignancies with less than a 2 year disease free interval at the time of dosing. Patients with adequately treated basal or squamous cell carcinoma of the skin, carcinoma in situ of the cervix or Stage A low-grade prostate cancer may enroll irrespective of the time of diagnosis.
* Patients who are receiving concomitant chemotherapy, immunotherapy, radiotherapy, or investigational therapy. Radiotherapy for palliation of related bone metastases is permitted upon the agreement between the investigator and the ImmunoGen Medical Monitor and as long as radiation does not involve target lesions that are followed for drug treatment response evaluation.
* Patients with any severe concurrent disease or condition, which in the judgment of the Investigator, would make the patient inappropriate for study participation. The disease or condition include, but are not limited to, one or more of the following: bleeding diathesis, uncontrolled chronic kidney or liver disease, uncontrolled diabetes, history of cardiac disease, myocardial infarction within the past 6 months, congestive heart failure, unstable angina pectoris, cardiac arrhythmia, and uncontrolled hypertension.
* Patients who must use contact lenses and cannot discontinue use of their contact lenses during the course of the clinical study. Patients must discontinue use of contact lenses prior to receiving study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-05; Primary Completion 2010-05 (Estimated); Study Completion 2010-09 (Estimated)

PRIMARY OUTCOMES:
response rate | year

SECONDARY OUTCOMES:
duration of response | as necessary
progression free survival | as necessary
safety and tolerability | while on study
Pharmacokinetic (PK) assessment | while on study
effect of huC242-DM4 on tumor uptake of FDG | while on study

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - UAB Comprehensive Cancer Center, Birmingham, Alabama
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - U.T. M.D. Anderson Cancer Center, Houston, Texas
  - South Texas Accelerated Research Therapeutics, San Antonio, Texas